CLINICAL TRIAL: NCT07071987
Title: A Multicenter, Randomized Controlled Trial to Evaluate the Efficacy of Thread Embedding Acupuncture in Reducing Postoperative Ileus After Colorectal Cancer Surgery
Brief Title: Effect of Thread Embedding Acupuncture on Postoperative Ileus Recovery After Colorectal Cancer Surgery: A Multicenter Randomized Controlled Trial
Acronym: THREAD-POI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: northernjiangsu008; 82373014 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-07-16; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Postoperative Ileus; LARS - Low Anterior Resection Syndrome
MeSH Terms: conditions — Colorectal Neoplasms; Low Anterior Resection Syndrome | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were blinded to their group assignment. In the sham group, blunt needles were placed at the same acupoints using adhesive pads without skin penetration or electrical stimulation, simulating the appearance of real thread embedding. Outcome assessors and investigators responsible for data collection and analysis were also blinded to the group allocation. Care providers performing the procedure were not blinded due to the nature of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thread embedding+Electroacupuncture Group (Experimental): Thread embedding at bilateral ST36, ST37, and PC6 at 2h after surgery and Electroacupuncture at same location at 2h, 24h, 48h, and 72h postoperatively
  Interventions: Procedure: Thread Embedding Acupuncture+Electroacupuncture
- Electroacupuncture Group (Other): Electroacupuncture
  Interventions: Procedure: Electroacupuncture
- Control Group (No Intervention): Standard perioperative management without any acupuncture-related intervention

INTERVENTIONS:
Procedure: Thread Embedding Acupuncture+Electroacupuncture — Thread embedding acupuncture will be administered at bilateral ST36, ST37, and PC6 acupoints at 2h after surgery and electroacupuncture at same acupoints at 2h 24h, 48h, and 72h after surgery. Absorbable polydioxanone sutures will be embedded into subcutaneous tissue using sterile embedding needles. All procedures will be conducted by licensed acupuncturists following standardized operating protocols.
  Arms: Thread embedding+Electroacupuncture Group
Procedure: Electroacupuncture — Electroacupuncture will be performed at the same bilateral acupoints (ST36, ST37, and PC6)
  Arms: Electroacupuncture Group

SUMMARY:
This multicenter, randomized, controlled trial aims to evaluate the efficacy and safety of thread embedding acupuncture (TEA) in promoting gastrointestinal recovery after laparoscopic colorectal cancer surgery. The primary outcome is the time to first flatus. Secondary outcomes include time to first defecation, tolerance to oral intake, length of hospital stay, and patient-reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years Diagnosed with stage I-III colorectal cancer Scheduled for elective laparoscopic colorectal resection ASA Physical Status I-III Ability to provide informed consent

Exclusion Criteria:

History of prior major abdominal surgery Emergency or palliative surgery Combined organ resection or open conversion Severe postoperative complications (e.g., anastomotic leak, GI bleeding) Severe cardiac, hepatic, renal, or psychiatric comorbidities Refusal to undergo acupuncture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to First Flatus | Up to 96 hours after surgery
  Time (in hours) from the end of surgery to the first passage of gas per rectum

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No